CLINICAL TRIAL: NCT01096823
Title: Iyengar Yoga for Young People With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lonnie Zeltzer, Distinguished Professor of Pediatrics, Anesthesiology, Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AR057318-01 (NIH)
Record Dates: First submitted 2010-03-24; First posted 2010-03-31 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Yoga; Adolescents; Young Adults
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iyengar Yoga (Experimental)
  Interventions: Behavioral: Iyengar Yoga
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: Iyengar Yoga — Iyengar Yoga classes twice a week for six weeks
  Arms: Iyengar Yoga

SUMMARY:
The purpose of this study is to compare a standardized 6 week Iyengar Yoga program (IYP) for adolescents and young adults with rheumatoid arthritis to a standard care wait-list condition. In addition to effects on function and pain, this study will explore intervention effects on disease activity, immune response, HRQOL, functionality, and mood. Results will shed light on the feasibility and potential efficacy of a novel intervention (Iyengar yoga) for rheumatoid arthritis symptoms.

The hypotheses are:

1. The IYP will be safe, acceptable and feasible: at least 80% of subjects will complete the IYP.
2. Following the IYP, participants will show significantly improved disease status, general functioning, arthritis-functioning and HRQOL relative to controls. The benefits will be apparent post-treatment and at two-month follow-up.
3. Following the IYP, participants will report significantly improved pain, immune response and mood compared to controls. These improvements will be evident at both post-treatment and at two-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* People with rheumatoid arthritis between the ages of 16-35
* Diagnosis of RA, according to the revised 1987 ACR criteria, or juvenile idiopathic arthritis (JIA) for at least 6 months
* Concomitant use of disease modifying antirheumatic medications (hydroxychloroquine, sulfasalazine, methotrexate, leflunomide, etc) biologic agents (infliximab, etanercept, adalimumab, abatacept, rituximab, anakinra) is permitted provided that the dose(s) have been stable for 4 weeks prior to screening, and may reasonably be expected to remain on stable doses throughout the duration of the trial
* Concomitant use of non-steroidal anti-inflammatory drugs (NSAIDs) and low dose corticosteroids (e.g prednisone at doses of 10 /day prednisone or equivalent is permitted provided that the dose(s) have been stable for 4 weeks prior to screening, and may reasonably be expected to remain on stable doses throughout the duration of the trial
* Disease activity, as defined using a 28 joint count by > 5 tender joints, > 5 swollen joints, and one of the following: ESR > 28 mm/hour, CRP > 1.5 mg/dL, duration of a.m. stiffness > 45 minutes
* Ability to provide written informed consent
* Ability to speak and understand English

Exclusion Criteria:

* Intra-articular steroid injections within 4 weeks of screening
* Treatment with any investigational agent within 8 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion that might affect the interpretation of the results or render the patient at high risk from treatment complications
* Inability to comply with study and follow-up procedures
* Currently pregnant
* Inability to speak or understand English
* Any recent injury.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lonnie K Zeltzer, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Pediatric Pain Program Research Offices, Los Angeles, California, United States

REFERENCES:
- [Derived] Evans S, Cousins L, Tsao JC, Subramanian S, Sternlieb B, Zeltzer LK. A randomized controlled trial examining Iyengar yoga for young adults with rheumatoid arthritis: a study protocol. Trials. 2011 Jan 21;12:19. doi: 10.1186/1745-6215-12-19. PMID 21255431

RESULTS

PARTICIPANT FLOW:
Groups:
- Waitlist Control: Standard of care waitlist control group
Period: Overall Study
Arm/Group | Iyengar Yoga | Waitlist Control
Started | 14 | 16
Completed | 11 | 15
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iyengar Yoga | Waitlist Control | Total
Number analyzed (Participants) | 11 | 15 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (2.9) | 27.1 (4.2) | 28.3 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Health Related Quality of Life - Short Form-36 (SF-36)
Description: The Health Related Quality of Life - Short Form-36 (SF-36) is a generic core HRQOL measure yielding an 8-scale profile of functional health and well being. The SF-36 performs comparatively better than other HRQOL measures in terms of reliability, validity, lightness of respondent/administrative burden. It can be completed in 5-10 minutes and has been used with children as young as 10 years of age.
  Subscales - all ranges 0-100 with higher scores indicating increased quality of life Bodily Pain, 2 items General Health, 5 items Vitality, 4 items Mental Health, 5 items
Time Frame: post intervention (within 2 weeks of completing intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iyengar Yoga | Waitlist Control
Number analyzed (Participants) | 11 | 15
units on a scale
  Bodily Pain Sub-Scale | 59.1 (19.2) | 59.3 (26.4)
  General Health Sub-Scale | 60.1 (21.4) | 47.0 (16.7)
  Vitality Sub-Scale | 64.5 (12.3) | 37.7 (21.7)
  Mental Health Sub-Scale | 81.6 (6.9) | 67.8 (19.5)

2. Primary Outcome: Pain Disability Index (PDI)
Description: The PDI assess the impact of pain on ability to participate in basic life activities, including social activity, sexual behavior, self-care and life-support activity. The PDI has been used with patients as young as 15. Good internal reliability (α = .82) and validity have been reported. It takes less than 5 minutes to complete.
  7 items, total measure range: 0-70, higher scores = higher interference/disability
Time Frame: post intervention (within 2 weeks of completing intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iyengar Yoga | Waitlist Control
Number analyzed (Participants) | 11 | 15
units on a scale | 13.5 (14.5) | 15.4 (17.3)

3. Primary Outcome: Health Assessment Questionnaire (HAQ)
Description: Items include questions about dressing and grooming, rising, eating, walking, hygiene, reaching, grip and making activities. The HAQ is one of the most widely recognized measures of patient functioning, with acceptable reliability and validity. It has been used successfully with adolescents as young as 13 years of age
  Range: 0-100, lower scores indicate better health
Time Frame: post intervention (within 2 weeks of completing intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iyengar Yoga | Waitlist Control
Number analyzed (Participants) | 11 | 15
units on a scale | 31.5 (28.5) | 55.9 (31.5)

4. Primary Outcome: Disease Activity Scale (DAS)28
Description: is a combined index that measures disease activity in patients with RA and remains a more thorough, established alternative to standard medical exams. This index includes a 28 tender joint count, 28 swollen joint count, Erythrocyte Sedimentation Rate (ESR), and general health assessment using a visual analogue scale. The ESR indirectly measures inflammation in the body and involves collecting blood samples, which will be performed by a qualified phlebotomist.
  The DAS score is a complicated formula based on many factors so there are no set ranges, but the published standards are as follows:
  "A DAS28 score of higher than 5.1 is indicative of high disease activity, whereas a DAS28 below 3.2 indicates low disease activity. A patient is considered to be in remission if they have a DAS28 lower than 2.6." Source: DAS-Score.nl. Available at http://www.das-score.nl/www.das-score.nl/index.html. Accessed February 5, 2009.
Time Frame: post intervention (within 2 weeks of completing intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iyengar Yoga | Waitlist Control
Number analyzed (Participants) | 11 | 15
units on a scale | 3.3 (1.2) | 3.3 (1.6)

ADVERSE EVENTS:
Arm/Group | Iyengar Yoga | Waitlist Control
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15
Other Adverse Events (participants affected / at risk) | 0/11 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No